CLINICAL TRIAL: NCT01839110
Title: A Randomized, Double-blind, Placebo Controlled, Multi-center Study to Assess the Effect of Ranolazine on Outcomes in Subjects With Pulmonary Hypertension and Right Ventricular Dysfunction Accompanied by a Comparative Study of Cellular Metabolism in Subjects With Pulmonary Hypertension With and Without Right Ventricular Dysfunction
Brief Title: Targeting the Right Ventricle in Pulmonary Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: The Cardiovascular Medical Research and Education Fund (Other); Brigham and Women's Hospital (Other); University of Maryland (Other); Yale University (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 817785
Record Dates: First submitted 2013-04-17; First posted 2013-04-24 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; right ventricular function; ranolazine
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ranolazine (Active Comparator): Ranolazine at 500mg by mouth twice per day and after two weeks will increase to 1000mg by mouth twice per day
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo by mouth twice per day
  Interventions: Drug: Placebo
- Observational (No Intervention): Patients with pulmonary hypertension who have normal RV function (RVEF >=45%) will undergo same procedures in the observational arm but will not receive an intervention.

INTERVENTIONS:
Drug: Ranolazine — Ranolazine at 500mg by mouth twice per day and after two weeks will increase to 1000mg by mouth twice per day and continue for a total of 26 weeks.
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Placebo by mouth twice per day for a total of 26 weeks.
  Arms: Placebo

SUMMARY:
This study is looking to see if giving ranolazine to subjects on stable pulmonary hypertension specific therapies but with right ventricular dysfunction (RVEF <45%) would improve their outcome. This study is accompanied by a baseline comparison of the metabolic profiling/microRNA/iPS cells of subjects with and without right ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary hypertension based on one of the following criteria: Idiopathic pulmonary arterial hypertension, Familial pulmonary arterial hypertension, pulmonary hypertension associated with connective tissue disease, chronic thromboembolic pulmonary hypertension-nonsurgical/distal vessel disease or patients who are reluctant to go to surgery within a 6-month period and are willing to participate, simple congenital such as repaired atrial septal defect or ventricular septal defect or unrepaired small atrial septal defect or ventricular septal defect with persistent and out of proportion pulmonary arterial hypertension, group 3 patients who have a component of pulmonary arterial hypertension, pulmonary arterial hypertension caused by conditions affect the veins and small vessels of the lungs, sickle cell disease, group 5 pulmonary hypertension such as polycythemia vera, essential thrombocythemia, sarcoidosis, or vasculitis, or metabolic disorder.
* WHO functional class II, III, or IV
* Mean pulmonary artery pressure >25 mmHg at rest
* Pulmonary capillary wedge pressure or left ventricular end diastolic pressure < 15 mmHg
* Baseline 6-minute walk test distance > 50 meters
* Stable on baseline existing PH specific therapy for 12 weeks with no dosage change within 28 days prior to screening.

Exclusion Criteria:

* Previous treatment with or prior sensitivity to ranolazine
* Any family history of corrected QT interval prolongation, congenital long QT syndrome, or receiving drugs that prolong the corrected QT interval
* Parenchymal lung disease showing total lung capacity < 50% of predicted OR forced expiratory volume at one second/forced vital capacity < 50%
* Portal hypertension associated with liver disease
* Left sided heart disease including any of the following: moderate or greater aortic or mitral valve disease, Any left ventricle cardiomyopathy, Left ventricular systolic dysfunction defined as an ejection fraction < 50%, Symptomatic coronary artery disease
* Uncontrolled hypertension
* Uncontrolled diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Han, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
IPD available upon request

REFERENCES:
- [Derived] Han Y, Forfia PR, Vaidya A, Mazurek JA, Park MH, Ramani G, Chan SY, Waxman AB. Rationale and design of the ranolazine PH-RV study: a multicentred randomised and placebo-controlled study of ranolazine to improve RV function in patients with non-group 2 pulmonary hypertension. Open Heart. 2018 Feb 23;5(1):e000736. doi: 10.1136/openhrt-2017-000736. eCollection 2018. PMID 29531764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine | Placebo | Observational
Started | 7 | 6 | 9
Completed | 4 | 4 | 6
Not Completed | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Observational | Total
Number analyzed (Participants) | 7 | 6 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (19.7) | 57.7 (6.8) | 53.2 (17.9) | 54.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 6 | 13
  Male | 4 | 2 | 3 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Changes in Right Ventricular Ejection Fraction
Description: right ventricular ejection fraction by cardiac MRI
Time Frame: 6 months
Population: Completers
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Ranolazine | Placebo | Observational
Number analyzed (Participants) | 4 | 3 | 6
percentage | 5.8 (2.0) | -4.7 (3.2) | 0.49 (3.2)

ADVERSE EVENTS:
Time Frame: 7 months. 6 months of trial and adverse events are gathered for 30 additional days
Arm/Group | Ranolazine | Placebo | Observational
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/6 | 0/9
Other Adverse Events (participants affected / at risk) | 5/7 | 2/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=7) | Placebo (N=6) | Observational (N=9)
heart failure hospitalization (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=7) | Placebo (N=6) | Observational (N=6)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
hyponatremia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
face edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT01839110/Prot_SAP_000.pdf